CLINICAL TRIAL: NCT04697043
Title: The Survival Benefit of Local Surgery in Stage IV of Breast Cancer
Brief Title: The Benefit of Surgery in Stage IV of Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 964635
Record Dates: First submitted 2020-12-14; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer Stage IV
Keywords: Surgery; Breast Cancer; Stage IV
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Centralized randomization will take place immediately after the diagnosis of primary distant metastatic breast cancer, using computer-generated randomization. dominant location of distant metastases (bone, soft tissue (lymph nodes and subcutaneous metastases) and visceral metastases), hormonal receptor status (ER and/ or PR positive or both negative) and HER2Neu status (overexpression yes or no) will be recorded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- systemic therapy followed by surgery (Experimental): ُThe main intervention is surgery. After the diagnosis of primary distant metastatic breast cancer, patients will be randomly allocated into two groups: A. systemic therapy followed by surgery if the disease is not progressive; B. Systemic therapy Patient selection criteria
  The eligibility criteria for the study are:
  - primary distant metastatic breast cancer (M1); - an anticipated survival of at least 6 months; - a histologically proven diagnosis of the breast tumor; - a known hormonal and HER2Neu status; - TNM classification: T1-T3, resectable T4 status, and N0-N3; - performance status and comorbidity should allow surgery and/or systemic therapy; - age ≥ 18 years;- written informed consent.
  Interventions: Procedure: Systemic therapy followed by surgery if the disease is not progressive
- Systemic therapy (No Intervention): After the diagnosis of primary distant metastatic breast cancer, patients will be randomly allocated into two groups: A. systemic therapy followed by surgery if the disease is not progressive; B. Systemic therapy Patient selection criteria
  The eligibility criteria for the study are:
  - primary distant metastatic breast cancer (M1); - an anticipated survival of at least 6 months; - a histologically proven diagnosis of the breast tumor; - a known hormonal and HER2Neu status; - TNM classification: T1-T3, resectable T4 status, and N0-N3; - performance status and comorbidity should allow surgery and/or systemic therapy; - age ≥ 18 years;- written informed consent.

INTERVENTIONS:
Procedure: Systemic therapy followed by surgery if the disease is not progressive — Primary systemic therapy (PST) or neoadjuvant therapy is used in nonmetastatic breast cancer to treat systemic disease earlier, decrease tumor bulk ideally to a complete pathological response (pCR), and reduce the extent of surgery. The systemic therapy followed by surgery if the disease is not progressive.
  Arms: systemic therapy followed by surgery

SUMMARY:
Treatment of Metastatic Breast Cancer is not usually considered curative. Recent retrospective studies have demonstrated that resection of the breast tumor in patients with primary metastatic breast cancer is associated with a significant improvement of the prognosis. In all these aforementioned studies, the decision to perform surgery could have been influenced by favorable prognostic factors, such as younger age, the presence of only one metastatic site, or good response to systemic therapy. To rule out the impact of potential confounders, most studies adjusted for age, tumor size, number and sites of metastases and hormone receptor status. In addition, some studies also adjusted for comorbidity or surgical margins. For example, in the study of Bafford et al., the benefit of surgery seemed confined to patients operated upon before diagnosis of metastatic disease and there was no survival advantage in patients who received an operation of the breast tumor after the diagnosis of the metastatic disease had taken place. This phenomenon was referred to as the stage migration bias. In a study by Leung et al., the benefit from surgery disappeared in the multivariate analysis when taking into account the use of chemotherapy. Finally, in a study by Cady et al. coding errors in the retrospectively collected dataset were found to explain part of the survival advantage. 4Therefore, this randomized controlled trial (RCT) has been initiated.

In the literature, several retrospective studies noted that 35-60% of patients with metastatic cancer at the time of diagnosis received local treatment of primary lesions, which resulted in a positive impact on survival. However, an analysis of 16,023 patients presenting with stage IV disease and an intact primary tumor compared outcomes between patients having surgery of the primary tumor to negative margins or no surgery. In a multivariate analysis adjusting for known prognostic factors, surgery reduced the HR for death to 0.61 (95% CI = 0.58 to 0.65). Multiple other retrospective studies from single institutions, registries, and population-based cohorts have confirmed this initial observation, but it is uncertain whether these studies reflect a real benefit for surgery or consistent selection bias. Three prospective randomized trials are examining the role of surgery in patients presenting with stage IV disease and an intact primary tumor. While awaiting the results of these trials, it is not known precisely how or when to integrate such surgical management into a standard medical therapy for metastatic breast cancer or which patients, in particular, are most likely to benefit from such treatment. 1 The aim of this study is to investigate the effect of surgery of the primary tumor in breast cancer patients with distant metastatic disease at initial diagnosis. According to the controversies in previous studies design of a study with the least confounding factor to decrease the bias seems to be necessary.

DETAILED DESCRIPTION:
After the diagnosis of primary distant metastatic breast cancer, patients will be randomly allocated into two groups: A. systemic therapy followed by surgery if the disease is not progressive; B. Systemic therapy Patient selection criteria

The eligibility criteria for the study are:

- primary distant metastatic breast cancer (M1); - an anticipated survival of at least 6 months; - a histologically proven diagnosis of the breast tumor; - a known hormonal and HER2Neu status; - TNM classification: T1-T3, resectable T4 status, and N0-N3; - performance status and comorbidity should allow surgery and/or systemic therapy; - age ≥ 18 years;- written informed consent.

Exclusion criteria are:

- primary invasive breast cancer in the medical history; - another malignancy within the last 10 years, besides basal cell carcinoma of the skin or early-stage cervical cancer; - surgical treatment and/or radiotherapy of the breast tumor before randomization; - irresectable T4 breast tumor; - synchronous bilateral breast cancer.

Randomization Centralized randomization will take place immediately after the diagnosis of primary distant metastatic breast cancer, using computer-generated randomization. dominant location of distant metastases (bone, soft tissue (lymph nodes and subcutaneous metastases) and visceral metastases), hormonal receptor status (ER and/ or PR positive or both negative) and HER2Neu status (overexpression yes or no) will be recorded.

Settings and location The study is a randomized controlled trial, which will be conducted at Tehran University of medical sciences, imam Khomeini hospital Treatment options During the study patients can be treated with surgery of the primary tumor (depending on randomization), systemic therapy The different treatment modalities are described below. Patients who are randomized to upfront surgery of the breast tumor will receive a lumpectomy or mastectomy depending on patient and tumor characteristics. Both types of surgery may be conducted as long as the intention is complete resection of the primary tumor, which is defined as having succeeded in obtaining free resection margins for the invasive component. The choice to perform an axillary lymph node dissection is left to the discretion of the treating physician but is highly recommended if palpable and/or tumor positive lymph nodes in the axillary region are present. If patients are randomized for systemic therapy, they may still be candidates for surgery of the primary tumor. In the case of local progression, breast surgery is allowed at any time to gain local control. Surgery for this group is primarily indicated when the treating physician beliefs the tumor may cause wound problems in near future, despite the use of systemic therapy. Patients will be treated with systemic therapy according to the guidelines. The choice of initial chemotherapy, immunotherapy, and endocrine therapy depends-among others-on ER and PR and HER2Neu status, dominant site of distant metastases, age, performance status, and comorbidity; but may also depend on the chance to reach a complete remission for example in minimal metastatic disease. In patients with a hormone receptor-positive tumor, hormonal treatment is indicated. In the case of rapid progression, chemotherapy is the treatment of choice. In HER2Neu positive disease and the use of an aromatase inhibitor, it is possible to add HER2Neu targeted therapy. Chemotherapy is offered to patients with hormone receptor-negative status, with extensive and fast-growing visceral metastases. For this study, we advise using at least an anthracycline, a taxane, and cyclophosphamide for the first 2-3 lines of treatment, if necessary in combination with targeted therapy, such as HER2- Neu targeted therapy, according to local practice.

Primary and secondary outcome measures The primary endpoint is the two-year survival. This is defined as the percentage of patients who survive two years after randomization. Secondary endpoints are quality of life, overall survival, number of unplanned local therapies, i.e. surgery or radiotherapy, number of axillary lymph node dissections or axillary radiotherapy, determination of pathological resection margin (margin status) in patients treated by surgery of the primary tumor.

Statistics Sample size calculation We are planning a randomized controlled trial with an equal number of patients in both treatment arms, an accrual interval of 36 months. Sample size calculation

Step 1: Calculation of the number of events with the following formula:

α=0.05 zα/2= 1.96 β=0.20 Zβ=0.84 π1=π2= 1/2: Equal allocation HR =0.50 Event =66

Step2: Calculation of the number of Patients with the following formula:

In this step, we assume the 40% of patients will die during the 2-years follow-up of the study. So the total number of desired patients will be 212. Therefore we need 106 patients in each group. Considering a 10% loss of patients, we should enter 118 patients in each group.

Following calculations were conducted:

Follow-up period= 2 years Suppose Incidence Rate (IR) = 25 events/person-2 years λt=0.5 at t= 2-year S(t)= exp{-λt}= exp{0.5}=0.60 1-0.60= 0.40 It means 40% of patients will die during 2 years of follow-up.

S1(2)= exp{-0.5}=0.60 S2(2)=exp (-0.5* HR}=0.78 Pr {event} = 1- {(0.60+0.78)/2}=0.31 N= 66/0.31=212 Total number n=106 each group

Number after considering 10% loss =118 /group

Data analysis Investigators will enter the information required by the protocol into the Case Report Forms (CRFs). The data from all investigators will be pooled and summarized with respect to demographic and baseline characteristics and efficacy and safety observations. Data will be presented for the complete intent-to-treat population. The primary endpoint will be analyzed in a Cox regression model, with the minimization factors as covariables. Interim analysis

ELIGIBILITY:
Inclusion Criteria:

Primary confirmed distant metastatic breast cancer (M1); A histologically proven diagnosis of the breast tumor; A known hormonal and HER2Neu status; Having TNM classification: T1-T3, resectable T4 status, and N0-N3; - performance status and comorbidity should allow surgery and/or systemic therapy; Accepting the surgery by written informed consent.

Exclusion criteria are:

No confirmed primary invasive breast cancer in the medical history Having another malignancy within the last 10 years, besides basal cell carcinoma of the skin or early-stage cervical cancer Having the history of surgical treatment and/or radiotherapy of the breast tumor before randomization Having irresectable T4 breast tumor Having synchronous bilateral breast cancer.

-

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 212 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-11-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
The number of participants with no more tumor in their body | from 6 months after surgery to 5 years
  Patients get rid of cancer and no more tumor in their body, no grows of tumor size.
  Treatment effect
PFS (progression free survival) | from 6 months after surgery to 5 years
  Patients be alive with no cancer
Overall Survival (OS) | from 6 months after surgery to 5 years
  Patients survival

SECONDARY OUTCOMES:
The number of participants with no more distant metastasis | from 6 months after surgery to 5 years
  No more distance metastasis and more than that the tumor regression

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran University of Medical Sciences, Tehran, Iran